CLINICAL TRIAL: NCT05293652
Title: Effect of Hydrocortisone Iontophoresis Versus Hydrocortisone Phonophoresis On Post Surgical Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elnaser Abd Elfattah Ghareeb, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Phd_mghareeb
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Scar; Hydrocortisone; Iontophoresis; Phonophoresis
MeSH Terms: conditions — Cicatrix | interventions — Iontophoresis; Phonophoresis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iontophosresis group (Experimental)
  Interventions: Other: Iontophoresis; Other: traditional PT program
- Phonophoresis group (Experimental)
  Interventions: Other: Phonophoresis; Other: traditional PT program
- Traditional group (Experimental)
  Interventions: Other: traditional PT program

INTERVENTIONS:
Other: Iontophoresis — Hydrocortisone iontophoresis
  Arms: Iontophosresis group
Other: Phonophoresis — Hydrocortisone Phonophoresis
  Arms: Phonophoresis group
Other: traditional PT program — Ultrasound and deep friction massage

SUMMARY:
The purpose of this study will be to compare the effect of hydrocortisone iontophoresis and hydrocortisone phonophoresis on the treatment of surgical scar and overall scar appearance.

DETAILED DESCRIPTION:
Scar contractures develop and extend to the underlying connective tissue and then muscles, leading to reduction in joint range of motion and affecting the day-to-day activities.

Most patients (irrespective of age, gender and ethnicity) believe that even a small improvement in scarring is worthwhile , any research that may help improve scar outcome is meaningful.

The need of this study has developed from the rarity of information about the difference between the effectiveness of iontophoresis and phonophoresis in enhancing the overall appearance of surgical scar.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* same approach of medications
* scar size varies from 5-15 cm

Exclusion Criteria:

* have cardiac / pacemakers
* have significant health problems
* obese patients (BMI more than 30)
* uncooperative patients

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Scar pliability | at baseline and after 3 months of intervention
  assessment of change in Scar pliability by using tonometer device

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelnaser, Assistant lecturer, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Horus University, Egypt, Damietta, Egypt